CLINICAL TRIAL: NCT06616324
Title: Virtual Reality: An Innovative Approach to Reduce Pain and Anxiety During Extracorporeal Shock Wave Lithotripsy - A Randomized Controlled Trial
Brief Title: Virtual Reality to Reduce Pain and Anxiety During Extracorporeal Shock Wave Lithotripsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMN-2024-06741
Record Dates: First submitted 2024-08-20; First posted 2024-09-27 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Pain; Virtual Reality; Lithotripsy
Keywords: Virtual Reality; Pain; Anxiety; VR; ESWL; Extracorporeal Shock Wave Lithotripsy; Lithotripsy; Non-pharmacological
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Due to the nature of VR, it is impossible to mask the patients and the healthcare providers administering the shockwave treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Standard treatment with Virtual Reality headset and Active-Noise-Cancelling headphones
  Interventions: Device: Virtual Reality
- Control Group (No Intervention): Standard treatment without VR headset and ANC-headphones

INTERVENTIONS:
Device: Virtual Reality — Participants in the intervention group will undergo ESWL according to standard treatment but with the addition of Virtual Reality and ANC-headphones as a supplement.
  Arms: Intervention

SUMMARY:
The objective of this study is to evaluate the impact of intraprocedural Virtual Reality (VR) as a non-pharmacological intervention for mitigating anxiety and pain during Extracorporeal Shock Wave Lithotripsy (ESWL). The hypothesis is that VR can effectively reduce both pain and anxiety levels in patients by diverting their cognitive focus, potentially leading to a decrease in pharmacological intervention requirements.

The primary outcome is pain at energy level 900 during ESWL for the intervention and the control group.

The secondary outcomes are as follows:

* Type and dose of analgesia
* Conductance scores/values
* Anxiety levels
* Patient satisfaction
* Procedure duration
* Adverse events

Participants will be randomized into either the intervention or control group. Both groups will undergo ESWL according to standard treatment; however, the intervention group will wear a Virtual Reality headset and noise-cancelling headphones during the procedure, while the control group will not

DETAILED DESCRIPTION:
The objective of this study is to evaluate the impact of intraprocedural Virtual Reality (VR) as a non-pharmacological intervention for mitigating anxiety and pain during Extracorporeal Shockwave Lithotripsy (ESWL). The hypothesis is that VR can effectively reduce both pain and anxiety levels in patients by diverting their cognitive focus, potentially leading to a decrease in pharmacological intervention requirements.

Furthermore, the study aims to gather data on patients' perspectives regarding the functionality and efficacy of VR technology in enhancing their intraprocedural experience. This includes an evaluation of VR's role in contribution to the overall procedural experience.

Introduction: According to the European Association of Urology (EAU) guidelines, urolithiasis is treated with ESWL, Ureteroscopy (URS), Percutaneous Nephrolithotomy (PNL), or other surgical treatments that may relieve the obstructive symptoms of the urinary tract. EAU recommends ESWL as the primary treatment for renal pelvic and proximal ureteral stones of <20 mm. The success of ESWL is closely related to factors such as the experience of the urologist using the machine, localization of the stone, urinary system anatomy, and the patient's compliance with the procedure. To ensure compliance, it is important to minimize patients' pain and anxiety. To handle pain and anxiety, various ways including both pharmacological and non-pharmacological approaches are in use today. Pharmacological control of pain and anxiety, including the use of sedation, is a complex decision that consider both benefits and potential risks. While not highly recommended due to the side effects associated with these agents, such as hypotension, respiratory depression, confusion, and limitations in ability to operate machines, sedation medication can be an effective means of managing pain and anxiety when used judiciously.

Non-pharmacological alternatives have been recommended for decreasing pain and anxiety during ESWL, as for example music which have been found beneficial in several studies. VR can immerse patients into a virtual environment and distract patients from e.g., unpleasant sounds, sights, and feelings. Integrating VR into hospital settings, has shown the potential to offer several advantages, such as promoting patients' distraction, knowledge, and information. The advantage lies in the engagement of multiple sensory perceptions, including hearing and vision, which can be beneficial in enhancing the potential for reduced experiences of pain and anxiety, as these perceptions typically strengthen humans' cognitive memory. The hypothesis is that distraction from VR can lower pain perception and reduce anxiety for patient undergoing EWSL compared with standard care.

Virtual Reality (VR) has been widely used in psychiatry and for children when they need to have a peripheral venous catheter inserted. Many studies show that VR has a distracting effect, and this distraction can be used to reduce both pain and anxiety. The novelty of this research study lies in using VR during ESWL so that the patient experiences less pain and anxiety. There is only one study from 2023, conducted in Belgium, which investigates whether VR is effective in reducing pain in kidney stone patients during ESWL. This study is a randomized controlled trial (RCT), and its results support the use of VR as a method for pain relief during ESWL.

There is a significant need for more evidence-based research studies in this area. With more research, it will be possible to better assess whether VR has the desired effect and relevance within medical procedures.

Method: The trial will be designed as a randomized controlled clinical trial while being adequately powered for the primary outcome. The randomization will be computer-generated randomization by the statistic programme R studio with sequence 1:1 by a colleague not associated to the study. The sample size estimation showed that 72 participants are needed with a 15% drop rate. The participants will be randomized into one of two groups. There will be randomization on the day of inclusion by REDcap which also store the data about the patients.

Because of VR's nature, it is impossible to blind the participants. The outcome assessors, investigators, data analysts, and manuscript writers will be blinded. The participants are patients undergoing urological procedure at Zealand University Hospital, Roskilde. All ASA scores are accepted.

All patients scheduled for ESWL will be screened based on the inclusion and exclusion criteria. Patients are eligible if they meet all inclusion criteria and none of the exclusion criteria. Intervention Group: Patients will receive ESWL using the EDAP-TMS model Sonolith i-sys machine with standard medication, supplemented by a Virtual Reality headset and Active-Noise-Cancelling (ANC) headphones, which will play a video of the patient's choice. Control Group: Patients will receive ESWL with standard medication, without the addition of VR or ANC-headphones. Participation in this trial will not result in prolonged admission or require additional follow-up visits.

The four different videos of what the patient can choose from, are developed specific for intraprocedural use and have been established in cooperation with people older than 65 years of age, private company Khora and Zealand University Hospital, Denmark and Lund University. The videos are created to fit different personalities and needs when persons undergo painful procedures. The development of the videos has focused on comprehending videos that have movement, colours, sound and pixels quality to prevent cyber sickness.

Standard intraprocedural management: All patients will follow the traditional standard treatment which includes Paracetamol and Ibuprofen as premedication with the possibility of receiving sublingual fentanyl during procedure to comfort the patient.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for ESWL at Region Zealand
* Age of 18 or above
* Ability to understand the trial protocol, risks, and benefits and provide signed informed consent

Exclusion Criteria:

* Inability to read and understand Danish.
* Uncooperativeness (as judged by investigators)
* Claustrophobia or fear of small spaces
* Disorders that prevent the person from wearing a VR device
* Highly visually or auditive impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain at energy level 900 | The outcome measure will be assessed from the start of the patient's ESWL treatment until the end of the procedure, with an average treatment duration of approximately 45 minutes.
  Data about the pain is registered at energy level 900 during the ESWL treatment for the intervention and the control group. The pain is measured by using the Numeric Rating Scale rating from 0-10. Zero is no pain at all and 10 is the worst imaginable pain. The outcome measure will be assessed during the patient ESWL treatment when the energy level of 900 is reached.

SECONDARY OUTCOMES:
Patient Satisfaction | The outcome measure will be assessed by the patient 1 hour or less after the ESWL treatment have ended.
  Patient satisfaction will be measured using a Likert scale from 1 to 5, where 1 and 2 indicate dissatisfaction, 3 is neutral, and 4 or 5 indicate satisfaction.
Adverse events | The outcome measure will be noted during or less than 1 hour after the ESWL treatment is finished.
  Adverse events are defined as any unwanted event, sign, or symptom occurring during the trial, whether the adverse is related to the VR head-mounted display or not.
  If any adverse events occur they will be noted.
Procedure duration | Measurements will be recorded for each individual during the treatment approximately 45 minutes.
  The procedure time will be recorded and is defined as the duration from the first shock wave to the last.
Pre- and intraprocedural pain | Measurements will be taken at the day for treatment for each individual. At arrival at preperations room and during the patients ESWL treatment approximately 2 hours time frame..
  Pain will be measured using the Numeric Rating Scale, rating from 0 to 10, where 0 represents no pain at all and 10 represents the worst imaginable pain. A lower score is favorable.
Anxiety | Measurements will be taken at the day for treatment for each individual. At arrival at preperations room and during the patients ESWL treatment approximately 2 hours time frame.
  Anxiety will be measured by using Numeric Rating Scale scale 0-10. Zero is no anxiety at all, and 10 is the worst imaginable anxiety. A lower score is favorable. To measure a more objective anxiety digital biomarkers by a proven wrist band made by Empatica will be used.
Conductance score/values | The outcome measure will be assessed from the start of the patient's ESWL treatment until the end of the procedure, with an average treatment duration of approximately 45 minutes.
  A machine that measures pain by monitoring the skin conductance. The PMD-200 uses a model based on skin conductance and other physiologic and hemodynamic changes and gives a Nociception Level Index (NOL) (20) from 0 to 100, where above 25 means treatment/pain medication is suggested. Therefore a score lower than 25 is favorable. The MedStorm PainSensor is a skin conductance algesimeter (SCA) that counts the peaks per second of skin conductance (when sympathetic nerves fire). A value over 0.06 suggests the level of nociception should be treated with pain medication(s). Therefore a score lower than 0.06 is favorable.
  Both machines will be used.
Type and dose of analgesia | The outcome measure will be assessed from the start of the patient's ESWL treatment until the end of the procedure, with an average treatment duration of approximately 45 minutes.
  Cumulative analgesia is the total amount of analgesia administrated before (at the same day) and during the procedure, and all analgetic medications will be collected for comparison. Different opioids will be converted to morphine IV equivalents for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Karsten L Lassen, PhD student, Principal Investigator — Urologisk Afdeling, Region Sjælland
Locations (1):
- Urologisk Afdeling, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang L, Zhang X, Pu Y, Zhang Y, Fan J. Global, Regional, and National Burden of Urolithiasis from 1990 to 2019: A Systematic Analysis for the Global Burden of Disease Study 2019. Clin Epidemiol. 2022 Aug 15;14:971-983. doi: 10.2147/CLEP.S370591. eCollection 2022. PMID 35996396
- [Background] Turk C, Petrik A, Sarica K, Seitz C, Skolarikos A, Straub M, Knoll T. EAU Guidelines on Diagnosis and Conservative Management of Urolithiasis. Eur Urol. 2016 Mar;69(3):468-74. doi: 10.1016/j.eururo.2015.07.040. Epub 2015 Aug 28. PMID 26318710
- [Background] Marsdin E, Noble JG, Reynard JM, Turney BW. Audiovisual distraction reduces pain perception during shockwave lithotripsy. J Endourol. 2012 May;26(5):531-4. doi: 10.1089/end.2011.0430. Epub 2012 Feb 8. PMID 22098167
- [Background] Ozsaker E, Diramali A. The effect of transcutaneous electrical nerve stimulation for pain relief during extracorporeal shock-wave lithotripsy procedure. Pain Manag Nurs. 2014 Mar;15(1):59-68. doi: 10.1016/j.pmn.2012.06.003. Epub 2012 Aug 18. PMID 24602425
- [Background] Yilmaz E, Ozcan S, Basar M, Basar H, Batislam E, Ferhat M. Music decreases anxiety and provides sedation in extracorporeal shock wave lithotripsy. Urology. 2003 Feb;61(2):282-6. doi: 10.1016/s0090-4295(02)02375-0. PMID 12597931
- [Background] Nakahara H, Furuya S, Masuko T, Francis PR, Kinoshita H. Performing music can induce greater modulation of emotion-related psychophysiological responses than listening to music. Int J Psychophysiol. 2011 Sep;81(3):152-8. doi: 10.1016/j.ijpsycho.2011.06.003. Epub 2011 Jun 24. PMID 21704661
- [Background] McCaffery M. Nursing approaches to nonpharmacological pain control. Int J Nurs Stud. 1990;27(1):1-5. doi: 10.1016/0020-7489(90)90018-e. PMID 2179151
- [Background] Cakmak O, Cimen S, Tarhan H, Ekin RG, Akarken I, Ulker V, Celik O, Yucel C, Kisa E, Ergani B, Cetin T, Kozacioglu Z. Listening to music during shock wave lithotripsy decreases anxiety, pain, and dissatisfaction : A randomized controlled study. Wien Klin Wochenschr. 2017 Oct;129(19-20):687-691. doi: 10.1007/s00508-017-1212-0. Epub 2017 May 17. PMID 28516381
- [Background] Wang Z, Feng D, Wei W. Impact of music on anxiety and pain control during extracorporeal shockwave lithotripsy: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2021 Jan 29;100(4):e23684. doi: 10.1097/MD.0000000000023684. PMID 33530169
- [Background] Weynants L, Chys B, D'hulst P, Merckx L, Van Besien J, Tailly T. Virtual reality for pain control during shock wave lithotripsy: a randomized controlled study. World J Urol. 2023 Feb;41(2):589-594. doi: 10.1007/s00345-023-04280-8. Epub 2023 Jan 21. PMID 36680576